CLINICAL TRIAL: NCT06503328
Title: Role of Specific microRNAs in Cluster Headache: Implications for Disease Phenotype and Neuropeptide Expression
Brief Title: Role of Specific microRNAs in Cluster Headache
Acronym: 5*1000
Status: Recruiting | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: miRNA - CH
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Cluster Headache
Keywords: MicroRNA; miR-34a-5p; miR-155; miR-382-5p; Peripheral blood mononuclear cells; CGRP; PACAP; VIP; Headache; Migraine
MeSH Terms: conditions — Cluster Headache; Headache; Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Controls: Healthy subjects without present or past history of headache according to ICHD-III criteria.
- Episodic Cluster Headache: Patients with a diagnosis of "3.1.1 Episodic Cluster Headache", according to ICHD-III criteria.
- Chronic Cluster Headache: Patients with a diagnosis of "3.1.2 Chronic Cluster Headache", according to ICHD-III criteria.

SUMMARY:
Cluster headache (CH) is a primary headache included in the trigeminal autonomic cephalalgias (TACs) according to the International Calssification of Headache Disorder, Third Edition. CH is characterized by a multifaceted and incompletely understood pathophysiology. Recent experimental evidence has increasingly emphasized the role of specific microRNAs (miRNAs) in the pathophysiology of primary headaches, including migraine.

In a recent study, we observed an upregulation in the gene expression of two miRNAs, miR-382-5p and miR-34a-5p, in peripheral blood mononuclear cells (PBMCs) of subjects with chronic migraine (CM). These miRNAs are involved in inflammation modulation and the release of γ-aminobutyric acid (GABA). Notably, this upregulation correlated with the migraine phenotype and its severity.

Several neuropeptides have been established to play an active role in CH. Studies by the Danish group have demonstrated that intravenous administration of CGRP, PACAP, or VIP can induce CH attacks in at least 50% of participants in the active phase of the disease.

However, no data currently exists regarding the potential involvement of miRNAs in CH. Given this context, the primary aim of this study is to investigate the gene expression of specific miRNAs (miR-382-5p, miR-34a-5p, and miR-155) in PBMCs and plasma levels of neuropeptides (CGRP, PACAP, VIP) in subjects with episodic CH in the active phase (eCH-act), episodic CH in the remission phase (eCH-rem), chronic CH (cCH), and healthy control subjects (HCs).

DETAILED DESCRIPTION:
Background Cluster headache (CH) is a primary headache included in the trigeminal autonomic cephalalgias (TACs) according to the International Calssification of Headache Disorder, Third Edition. CH is characterized by a multifaceted and incompletely understood pathophysiology. The hypothalamus, the trigeminal-vascular complex, and the trigeminal-autonomic reflex are believed to play a significant role.

Increasing experimental evidence has highlighted the involvement of specific microRNAs (miRNAs) in the chronic pain and primary headaches, including migraine. miRNAs are small endogenous noncoding RNAs that are around 22 nucleotides in length. miRNAs operate as post-transcriptional regulator of gene expression by promoting messenger RNA (mRNA) degradation or repressing mRNA translation. The regulation process performed by miRNAs is complex and articulated since an individual miRNA might target hundreds of different mRNAs, and conversely, each mRNA may be regulated by multiple miRNAs. It has been estimated that more than 60% of all protein-coding genes are regulated by miRNAs which consequentially determine the pleiotropic modulation of a wide variety of cellular processes involving differentiation, development and signaling. miRNAs are involved in the generation and maintenance of pain and several evidence suggest that specific miRNAs could play a role in migraine.

In a recent study, we observed an upregulation of gene expression in two miRNAs, miR-382-5p and miR-34a-5p, in peripheral blood mononuclear cells (PBMCs) in subjects with chronic migraine (CM). These miRNAs are involved in inflammation modulation and the release of γ-aminobutyric acid (GABA) compared to individuals with episodic migraine and healthy subjects (HCs). These findings underscore a correlation between the gene expression of these miRNAs and the migraine phenotype, as well as its severity.

Recent studies suggest an active role for certain neuropeptides in CH. The Danish group has indeed demonstrated that the intravenous administration of CGRP, PACAP, or VIP can induce acute CH attacks in at least 50% of participants when studied in the active phase of the disease.

As of now, there is no data regarding the potential involvement of miRNAs in CH. This study aims to provide a detailed exploration of the role of miRNAs in cluster headache, contributing to our understanding of the pathophysiology of this primary headache disorder. Furthermore, the results obtained may pave the way for the development of a new generation of molecules that could be used in the field of CH, such as miRNA agonists (Agomir) and antagonists (Antagomir).

Aims The primary objective of our current project is to investigate the peripheral expression of miRNAs implicated in pain modulation (miR-382-5p, miR-34a-5p, and miR-155) in subjects with episodic CH in the active phase (eCH-act), episodic CH in the remission phase (eCH-rem), chronic CH (cCH), and healthy control subjects (HC).

Methods

All subjects will perform a single evaluation over time during which they will undergo:

* explanation of study procedures and informed consent signing
* screening visit
* clinical and demographic data collection (based on revision of a headache diary)
* fasting venous blood sampling
* administration of questionnaires

All subjects will be evaluated in the morning, after night fasting. For subjects affected by cCH or eCH-act, sampling is expected to be carried out in the inter-critical phase, as defined by the absence of CH attacks for at least 3 hours in patients with eCH and for at least 8 hours in patients with cCH. After blood sampling, patients will stay at Center to complete a set of questionnaires. This will allow the investigator to monitor the patients for at least 2 hours, to exclude that a blood sampling is performed immediately before a CH attack.

For patients with eCH, the "active" and "remission" phases will be defined as follows:

* Active phase: the phase during which CH attacks have been present for at least 7 days.
* Remission phase: characterized by an absence of cluster headache attacks for at least 15 consecutive days without pharmacological therapy.

miR-382-5p, miR-34a-5p and miRNA-155 gene expression will be evaluated in PBMCs by real-time reverse transcription (RT-PCR). This assessment will be normalized with U6 (a type of small nuclear RNA used as housekeeping gene) and expressed as Relative Quantification (RQ). Plasma levels of CGRP alpha, PACAP and VIP will be measured using validated commercial ELISA kits. A detailed description of the methods planned for the biochemical analyses could be found here: https://doi.org/10.1186/s10194-020-01189-0.

The set of clinical questionnaires will include: Migraine Disability Assessment (MIDAS), Headache Impact Test (HIT-6), Cluster headache Impact Questionnarie (CHIQ).

Sample size calculation and pre-planned statistical analysis The following parameters were considered for the calculation: Effect Size: 0.5; alpha error: 0.05; beta error: 0.05 (power: 95%); number of groups: 4.

Sample size calculation was conducted using the freeware platform G*Power (ver. 3.1.9.7) for an ANOVA test with Bonferroni correction applied to the 4 groups. The minimum suggested sample size is 76 subjects (19 subjects per group). To account for potential variability, we plan to enroll a total of 100 subjects, with 25 subjects per group.

Parametric or non-parametric correlations will be used to measure the relationship between biochemical variables and clinical variables. Multivariate analyses will be performed according to the results of the univariate analysis. Statistical significance will be set at the 5% level (p<0.05).

ELIGIBILITY:
- Healthy Controls

Inclusion Criteria:

* age between >18 and <65 years

Exclusion Criteria:

* diagnosis of primary and/or secondary headache according to ICHD-III criteria (only diagnosis of sporadic tension type headache is allowed)
* diagnosis of neurological disorders
* diagnosis of medical conditions considered clinically relevant by the researcher
* pregnant and lactating women
* taking NSAIDs, triptans or opiates in the previous 24 hours
* Episodic Cluster Headache

Inclusion Criteria:

* diagnosis of Episodic Cluster Headache according to ICHD-III criteria (at least 1 year at screening)
* age between >18 and <65 years of both genders

Exclusion Criteria:

* concomitant diagnosis of other primary and/or secondary headache according to ICHD-III criteria (only diagnosis of sporadic tension headache is allowed)
* diagnosis of other neurological disorders
* diagnosis of medical conditions considered clinically relevant by the researcher
* diagnosis of chronic pain syndrome of any nature
* pregnant and lactating women
* use of substances of abuse
* Chronic Cluster Headache

Inclusion Criteria:

* diagnosis of Chronic Cluster Headache according to ICHD-III criteria (at least 1 year at screening)
* age between >18 and <65 years of both genders

Exclusion Criteria:

* concomitant diagnosis of other primary and/or secondary headache according to ICHD-III criteria (only diagnosis of sporadic tension headache is allowed)
* diagnosis of other neurological disorders
* diagnosis of medical conditions considered clinically relevant by the researcher
* diagnosis of chronic pain syndrome of any nature
* pregnant and lactating women
* use of substances of abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We aim to enroll a representative population of patients affected by eCH in the active phase and in the remission phases and cCH. All patients will be consecutively enrolled among those attending the clinics of the Headache Science Center of the IRCCS Mondino Foundation of Pavia (Italy).
  A set of healthy controls, without a present or past diagnosis primary or secondary headaches, will be enrolled as control group.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
PBMCs gene expression of miR-382-5p | Single evaluation at study visit - baseline (T0)
  miR-382-5p gene expression in PBMCs will be evaluated by real-time reverse transcription (RT-PCR). This assessment will be then normalized with U6 (a type of small nuclear RNA used as housekeeping gene) and expressed as Relative Quantification (RQ).

SECONDARY OUTCOMES:
PBMCs gene expression of miR-34a-5p and miR-155 | Single evaluation at study visit - baseline (T0)
  miR-34a-5p and miRNA-155 gene expression will be evaluated by real-time reverse transcription (RT-PCR). This assessment will be then normalized with U6 (a type of small nuclear RNA used as housekeeping gene) and expressed as Relative Quantification (RQ).
Plasma levels of CGRP alpha, PACAP and VIP | Single evaluation at study visit - baseline (T0)
  Plasma levels of CGRP alpha, CGRP beta, PACAP and VIP will be measured using validated commercial ELISA kits.
Score of MIDAS, HIT-6, and CHIQ | Single evaluation at study visit - baseline (T0)
  MIDAS, HIT-6, CHIQ represent validated clinical scales to rate CH related disability.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Mondino Foundation, Pavia, Italy

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Ahmad L, Demartini C, Corrado M, et al. Expression of Selected microRNAs in Migraine: A New Class of Possible Biomarkers of Disease? Processes 2021; 9: 2199.
- [Background] Greco R, De Icco R, Demartini C, Zanaboni AM, Tumelero E, Sances G, Allena M, Tassorelli C. Plasma levels of CGRP and expression of specific microRNAs in blood cells of episodic and chronic migraine subjects: towards the identification of a panel of peripheral biomarkers of migraine? J Headache Pain. 2020 Oct 16;21(1):122. doi: 10.1186/s10194-020-01189-0. PMID 33066724
- [Background] Welch KM, Chabi E, Bartosh K, Achar VS, Meyer JS. Cerebrospinal fluid gamma aminobutyric acid levels in migraine. Br Med J. 1975 Aug 30;3(5982):516-7. doi: 10.1136/bmj.3.5982.516. PMID 1164613
- [Background] Vollesen ALH, Snoer A, Beske RP, Guo S, Hoffmann J, Jensen RH, Ashina M. Effect of Infusion of Calcitonin Gene-Related Peptide on Cluster Headache Attacks: A Randomized Clinical Trial. JAMA Neurol. 2018 Oct 1;75(10):1187-1197. doi: 10.1001/jamaneurol.2018.1675. PMID 29987329
- [Background] Vollesen ALH, Snoer A, Chaudhry B, Petersen AS, Hagedorn A, Hoffmann J, Jensen RH, Ashina M. The effect of pituitary adenylate cyclase-activating peptide-38 and vasoactive intestinal peptide in cluster headache. Cephalalgia. 2020 Nov;40(13):1474-1488. doi: 10.1177/0333102420940689. Epub 2020 Sep 22. PMID 32962406
- [Background] Kadir RRA, Alwjwaj M, Bayraktutan U. MicroRNA: An Emerging Predictive, Diagnostic, Prognostic and Therapeutic Strategy in Ischaemic Stroke. Cell Mol Neurobiol. 2022 Jul;42(5):1301-1319. doi: 10.1007/s10571-020-01028-5. Epub 2020 Dec 24. PMID 33368054
- [Background] Gallardo VJ, Gomez-Galvan JB, Asskour L, Torres-Ferrus M, Alpuente A, Caronna E, Pozo-Rosich P. A study of differential microRNA expression profile in migraine: the microMIG exploratory study. J Headache Pain. 2023 Feb 17;24(1):11. doi: 10.1186/s10194-023-01542-z. PMID 36797674